CLINICAL TRIAL: NCT03699839
Title: Reducing the Burden of Influenza After Solid-Organ Transplantation: the STOP-FLU Trial [Swiss Trial in Solid Organ Transplantation on Prevention of Influenza]
Brief Title: Reducing the Burden of Influenza After Solid-Organ Transplantation
Acronym: STOP-FLU
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oriol Manuel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Bern (Other); University Hospital, Geneva (Other); University of Zurich (Other); Cantonal Hospital of St. Gallen (Other); Fondazione Epatocentro Ticino (Other); Cantonal Hospital Chur (Unknown); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor-Investigator, Oriol Manuel, Principal Investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-01922
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Influenza; Organ Transplantation
Keywords: Vaccination; Adjuvanted vaccine; High-dose vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- High dose influenza vaccine (Experimental): Administration of high-dose influenza vaccine
  Interventions: Biological: High-dose influenza vaccine
- MF59-adjuvanted influenza vaccine (Experimental): Administration of MF59-adjuvanted vaccine
  Interventions: Biological: MF59-adjuvanted influenza vaccine
- Standard influenza vaccine (Active Comparator): Administration of standard intramuscular influenza vaccine
  Interventions: Biological: Standard intramuscular influenza vaccine

INTERVENTIONS:
Biological: High-dose influenza vaccine — The experimental intervention consists in an intramuscular injection of a MF59-adjuvanted trivalent inactivated influenza vaccine containing 15 µg of antigen per strain (Fluad®) or an intramuscular injection of trivalent inactivated influenza vaccine containing 60 µg of antigen per strain (Fluzone-HD®) and will be performed at day 0.
  Arms: High dose influenza vaccine
Biological: MF59-adjuvanted influenza vaccine — The experimental intervention consists in an intramuscular injection of a MF59-adjuvanted trivalent inactivated influenza vaccine containing 15 µg of antigen per strain (Fluad®) or an intramuscular injection of trivalent inactivated influenza vaccine containing 60 µg of antigen per strain (Fluzone-HD®) and will be performed at day 0.
  Arms: MF59-adjuvanted influenza vaccine
Biological: Standard intramuscular influenza vaccine — The control intervention consists in an intramuscular injection of one dose of VaxigripTetra®, the standard non-adjuvanted intramuscular influenza vaccine (as routinely done).
  Arms: Standard influenza vaccine

SUMMARY:
Influenza is associated with significant morbidity and mortality in solid-organ transplant (SOT) recipients and it is mainly prevented by seasonal influenza vaccination. Unfortunately, the immunogenicity of standard influenza vaccine is suboptimal in this population. Vaccination with a high-dose (HD) influenza vaccine or an MF59-adjuvanted (MF59a) vaccine have significantly reduced the incidence of influenza and increased the immunogenicity of influenza vaccine in the elderly. The investigators will compare the immunogenicity and efficacy of two new vaccination strategies, consisting in vaccination with a HD influenza vaccine or an MF59a influenza vaccine, to the standard-dose non-adjuvanted vaccination (standard of care) in a population of SOT recipients.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to compare the immunogenicity of two novel vaccination strategies, consisting in vaccination with a HD influenza vaccine or an MF59a influenza vaccine, to the standard-dose non-adjuvanted vaccination (standard of care) in a population of SOT recipients.

The main secondary objectives are to evaluate the efficacy of the novel vaccination strategies in reducing the incidence of influenza, to correlate the humoral responses to vaccination with protection from influenza and to assess the influence of immunosuppression on influenza vaccine responses.

Safety objectives include the assessment of the reactogenicity of the different vaccines and to describe the incidence of acute rejection and the development of anti-Human Leucocyte Antigens (HLA) antibodies after vaccination.

Study design: Prospective double-blinded randomized controlled three-arm parallel group superiority multicenter trial.

Inclusion / Exclusion criteria: Study participants will be enrolled among ≥18-year old stable SOT recipients ≥3 months after transplantation, regularly followed at their respective outpatient clinic at the 7 transplant centers and scheduled to receive the annual influenza vaccine. Candidates will be excluded in case of previous severe reaction or allergy to one of the study vaccines or in case of treatment for acute rejection, among others.

Measurements and procedures: At day 0, after giving informed consent, eligible patients will be randomized in a 1:1:1 ratio into 3 arms: standard quadrivalent intramuscular vaccine (control), HD trivalent vaccine and MF59a trivalent vaccine. After vaccination participants will be followed for a period of 6 months. Safety will be assessed immediately after vaccination and 7, 28 and 180 days after vaccination, and blood sampling for immunogenicity analysis will be performed at baseline, 7, 28 and 180 days after vaccination. Additionally to evaluate the vaccine safety, anti-HLA antibodies will be measured at baseline and at days 28 and 180 after vaccination. Hemagglutinin titers will be determined by hemagglutination inhibition assay (HIA) according to standardized methods. During the influenza season, the development of influenza will be systematically assessed by polymerase chain reaction (PCR) by surveillance nasopharyngeal swab.

Study Product / Intervention: The study intervention consists in the intramuscular administration of either a HD vaccine (containing 60 µg of antigen of each of the three viral strains) [Fluzone-HD®] or a MF59a vaccine (containing 15 µg of antigen of each of the three viral strains with a MF59 adjuvant) [Fluad®].

Control Intervention: The control intervention consists in the administration of the standard quadrivalent non-adjuvanted intramuscular influenza vaccine (VaxigripTetra®), containing 15 µg of each of the four viral strains.

Number of Participants with Rationale: The investigators plan to enroll 780 patients (260 patients per study group). Sample size was calculated to find a significant difference between the three groups for the primary endpoint. The lowest seroconversion rate of 46% for standard dose, a mid seroconversion rate of 59% with MF59a vaccine, and the highest seroconversion rate of 70% with HD vaccine has been assumed. A 10% drop out rate is assumed and the number of patients has been rounded up to get balanced groups. In each group 260 patients are required which amounts to 780 patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent
* Age ≥18 years
* Stable outpatients based on clinical judgement
* ≥ 3 months after solid organ transplantation

Exclusion Criteria:

* Known hypersensitivity to any component (antigen, adjuvant, excipient or preservative) of study vaccines; the composition of the study vaccines is as follows:

  * VaxigripTetra®: hemagglutinin, egg protein, formaldehyde, octylphenol ethoxylate/octoxynol 9 (Triton® X-100), neomycin
  * Fluad®: hemagglutinin, neuraminidase, egg protein, squalene, polysorbate 80, sorbitan trioleate, sodium citrate, citric acid, kanamycin sulphate, neomycin sulphate, barium sulphate, formaldehyde, cetyl trimethylammonium bromide
  * Fluzone-HD®: hemagglutinin, egg protein, formaldehyde, octylphenol ethoxylate/octoxynol 9 (Triton® X-100)
* Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barré Syndrome)
* Ongoing therapy for rejection (including steroid pulse or prednisone > 2mg/kg/day over more than 14 days)
* Ongoing therapy with intravenous immunoglobulin (IVIG) and/or eculizumab
* Current or past (within 6 months) therapy with rituximab
* Abo incompatible transplantation
* Unable to comply with study protocol
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Vaccine response rate | day 28 after vaccination
  Seroconversion rate for at least one viral antigen

SECONDARY OUTCOMES:
Influenza infection | Within 6 month after vaccination
  PCR positive for influenza in a nasopharyngeal swab or other clinical specimen
Seroprotection rates | At day 28 and month 6 after vaccination
  Antibody levels >40 after vaccination
Reactogenicity | within 28 days after vaccination
  Self-collected adverse events
Development of anti-HLA antibodies | Within 6 months post vaccination
  De novo anti-HLA antibodies measured by Luminex

CONTACTS AND LOCATIONS:
Locations (9):
- Hospitales Universitarios Virgen del Rocio, Seville, Andalusia, Spain
- Switzerland (8):
  - Cantonal Hospital Chur, Chur, Kanton Graubünden
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Hopitaux Universitaires de Genève, Geneva
  - CHUV, Lausanne
  - Epatocentro Ticino, Lugano
  - Canton Hospital St-Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kumar D, Michaels MG, Morris MI, Green M, Avery RK, Liu C, Danziger-Isakov L, Stosor V, Estabrook M, Gantt S, Marr KA, Martin S, Silveira FP, Razonable RR, Allen UD, Levi ME, Lyon GM, Bell LE, Huprikar S, Patel G, Gregg KS, Pursell K, Helmersen D, Julian KG, Shiley K, Bono B, Dharnidharka VR, Alavi G, Kalpoe JS, Shoham S, Reid GE, Humar A; American Society of Transplantation H1N1 Collaborative Study Group. Outcomes from pandemic influenza A H1N1 infection in recipients of solid-organ transplants: a multicentre cohort study. Lancet Infect Dis. 2010 Aug;10(8):521-6. doi: 10.1016/S1473-3099(10)70133-X. Epub 2010 Jul 9. PMID 20620116
- [Result] Manuel O, Estabrook M; AST Infectious Diseases Community of Practice. RNA respiratory viruses in solid organ transplantation. Am J Transplant. 2013 Mar;13 Suppl 4(Suppl 4):212-9. doi: 10.1111/ajt.12113. No abstract available. PMID 23465014
- [Result] Mombelli M, Rettby N, Perreau M, Pascual M, Pantaleo G, Manuel O. Immunogenicity and safety of double versus standard dose of the seasonal influenza vaccine in solid-organ transplant recipients: A randomized controlled trial. Vaccine. 2018 Oct 1;36(41):6163-6169. doi: 10.1016/j.vaccine.2018.08.057. Epub 2018 Sep 1. PMID 30181045
- [Result] Kumar D, Campbell P, Hoschler K, Hidalgo L, Al-Dabbagh M, Wilson L, Humar A. Randomized Controlled Trial of Adjuvanted Versus Nonadjuvanted Influenza Vaccine in Kidney Transplant Recipients. Transplantation. 2016 Mar;100(3):662-9. doi: 10.1097/TP.0000000000000861. PMID 26335915
- [Result] Koller MT, van Delden C, Muller NJ, Baumann P, Lovis C, Marti HP, Fehr T, Binet I, De Geest S, Bucher HC, Meylan P, Pascual M, Steiger J. Design and methodology of the Swiss Transplant Cohort Study (STCS): a comprehensive prospective nationwide long-term follow-up cohort. Eur J Epidemiol. 2013 Apr;28(4):347-55. doi: 10.1007/s10654-012-9754-y. Epub 2013 Apr 2. PMID 23546766
- [Derived] Mombelli M, Neofytos D, Huynh-Do U, Sanchez-Cespedes J, Stampf S, Golshayan D, Dahdal S, Stirnimann G, Schnyder A, Garzoni C, Venzin RM, Magenta L, Schonenberger M, Walti L, Hirzel C, Munting A, Dickenmann M, Koller M, Aubert JD, Steiger J, Pascual M, Mueller TF, Schuurmans M, Berger C, Binet I, Villard J, Mueller NJ, Egli A, Cordero E, van Delden C, Manuel O. Immunogenicity of High-Dose Versus MF59-Adjuvanted Versus Standard Influenza Vaccine in Solid Organ Transplant Recipients: The Swiss/Spanish Trial in Solid Organ Transplantation on Prevention of Influenza (STOP-FLU Trial). Clin Infect Dis. 2024 Jan 25;78(1):48-56. doi: 10.1093/cid/ciad477. PMID 37584344